CLINICAL TRIAL: NCT04712825
Title: Effect of Medical Hypnosis in Virtual Reality on Insomnia Disorders: a Monocentric, Randomized, Open-label, Comparative Study.
Brief Title: Effect of Medical Hypnosis in Virtual Reality on Insomnia Disorders
Acronym: EMERITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HypnoVR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPNOVR-RIPH-2020-2
Record Dates: First submitted 2020-12-08; First posted 2021-01-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Insomnia Chronic
Keywords: Virtual reality; Hypnosis; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioural therapy (Active Comparator): Cognitive-behavioural therapy sessions
  Interventions: Behavioral: Cognitive-behavioural therapy
- Virtual Reality Hypnosis (Experimental): Virtual Reality Hypnosis sessions
  Interventions: Device: HypnoVR® device

INTERVENTIONS:
Behavioral: Cognitive-behavioural therapy — Cognitive-behavioural therapy sessions during 6 weeks of treatment
  Arms: Cognitive-behavioural therapy
Device: HypnoVR® device — HypnoVR® sessions during 6 weeks of treatment
  Arms: Virtual Reality Hypnosis

SUMMARY:
The prevalence of chronic insomnia is 13.3% in France in 2019 (8.9 million). The consequences for these people are multiple: drowsiness, memory problems, difficulty concentrating, anxiety.

Cognitive and Behavioral Therapy (CBT) is today the reference treatment recommended by the "Haute Autorité de Santé" and the American College of Physicians for chronic insomnia. Today, however, few patients use CBT treatment due to the lack of trained practitioners, the cost of non-reimbursed sessions and the time and involvement that these sessions require.

Several clinical trials have shown beneficial effects of hypnotherapy on sleep disorders. The hypothesis of this work is that the use of hypnosis in virtual reality improves sleep time in patients suffering from insomnia disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patient suffering from insomnia as defined in the Diagnostic and Statistical Manual of Mental Disorders V (DMS-V) and the International Classification of Sleep Disorders.

Exclusion Criteria:

1. Patient who, in the judgment of the investigator, has a disease that may preclude participation in study procedures.
2. Minor subject
3. Subject under judicial protection, guardianship or curatorship
4. Inability to give informed information about the subject: demented patients, psychotic patients or follow-up for a psychiatric pathology
5. Unbalanced epilepsy
6. Hearing and/or visual disorders that contraindicate the use of virtual reality headphones
7. Patient with a language barrier
8. Pregnant or breastfeeding patient
9. Subject in period of exclusion (determined by a previous or current study)
10. Patient Refusal
11. Patient currently being treated for depression, alcoholism or drug addiction.
12. Patient using drug treatment for insomnia not stabilized within 2 weeks prior to the start of the study.
13. Patient starting psychological, complementary or alternative medicine treatment for insomnia within 2 weeks prior to the start of the study, or during the study.
14. Patient receiving or having received CBT treatment for insomnia within the last 6 months.
15. Patient diagnosed with sleep apnea, involuntary limb movement, restless legs syndrome.
16. Patient with diagnosed medical conditions that cause insomnia: psychotic disorder, bipolar disorder, dementia, generalized anxiety disorder, panic disorder, manic disorder, schizophrenia, cancer.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Time to sleep | after 6 weeks of treatment
  Demonstrate a decrease in time to sleep after treatment, by polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- SELARL Respire, Haguenau, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR